CLINICAL TRIAL: NCT05098470
Title: Effects of Modulators of Gluconeogenesis, Glycogenolysis and Glucokinase Activity on Endogenous Glucose Production in Type 2 Diabetes
Brief Title: Effects of Modulators of Gluconeogenesis, Glycogenolysis and Glucokinase Activity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rita Basu, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 210395; R01DK029953 (NIH)
Record Dates: First submitted 2021-10-08; First posted 2021-10-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Insulin Glargine; Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Insulin Glargine (Active Comparator)
  Interventions: Drug: Insulin Glargine
- Dorzagliatin (Experimental)
  Interventions: Drug: Dorzagliatin

INTERVENTIONS:
Drug: Metformin — 1500-2000 mg per day for 8 weeks
  Arms: Metformin
Drug: Insulin Glargine — Long-acting insulin for 8 weeks
  Arms: Insulin Glargine
Drug: Dorzagliatin — Oral Glucokinase Activator 75 mg twice daily for 8 weeks
  Arms: Dorzagliatin

SUMMARY:
It has been shown that individuals with type 2 diabetes have higher blood sugar throughout the night than individuals without type 2 diabetes. However, it is still unknown if this rise in blood sugar can be controlled using medications.

This study will examine the effects of three different diabetes treatments to determine if they improve night time blood sugars. Participants will be randomly assigned for 8 weeks to one of the following three groups:

GROUP 1: Insulin. Participants will be instructed on self-injecting insulin glargine once-daily in the morning. The dose will be increased by the study team to avoid episodes of low blood sugar and to maintain fasting blood sugar concentrations between 70 to 180 mg/dl.

GROUP 2: Metformin. Participants will start the drug (500 mg twice daily) with meals. After 72 hours and in the absence of side effects, they will increase the dose to 500 mg with breakfast and 1,000 mg with supper. After a further 72 hours and in the absence of side effects, they will increase the dose to 1,000 mg twice daily with meals and continue until the end of the trial. The dose will be adjusted by the study team to maintain fasting blood sugar concentrations between 70 to 180 mg/dl.

GROUP 3: Dorzagliatin. This medication dose will be 75 mg twice daily. The investigators anticipate fasting glucose concentrations will be between 70 to 180 mg/dl since the dose of this medication cannot be titrated.

ELIGIBILITY:
Inclusion Criteria:

* BMI:25-40 kg/m2.
* HbA1C ≤ 9% on lifestyle therapy with or without monotherapy with metformin or sulphonylureas (SU); or combination therapies (metformin and SU, DPPIV inhibitors, only short acting GLP-1 analogues exenatide (Byeta) and liraglutide (Victoza).

Exclusion Criteria:

* Insulin therapy
* SGLT2 inhibitors
* Long acting GLP-1 analogues
* TZDs
* Medications affecting GI motility (e.g., erythromycin, pramlintide).
* Medications that may affect glucose metabolism such as corticosteroids, tricyclic-antidepressants, benzodiazepines, opiates, barbiturates, and anticoagulants.
* Unstable diabetic retinopathy, microalbuminuria, macrovascular disease.
* Upper GI disorder/surgery, debilitating chronic disease, anemia, and symptoms of undiagnosed illnesses.
* History of alcoholism or substance abuse.
* Pregnancy or breast feeding, or other comorbidities precluding participation.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Contribution of gluconeogenesis (GNG) to endogenous glucose production (EGP) | 8 weeks
  Ratio of GNG to total EGP

SECONDARY OUTCOMES:
Contribution of glycogenolysis (GLY) to EGP | 8 weeks
  Ratio of GLY to total EGP
Glucokinase activity | 8 weeks
  UDP glucose flux

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rita Basu, Birmingham, Alabama
  - University of Virginia, Charlottesville, Virginia

DOCUMENTS (1):
  • Informed Consent Form (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT05098470/ICF_000.pdf